CLINICAL TRIAL: NCT04302194
Title: Early Dietary Treated Patients With Phenylketonuria Can Achieve Normal Growth and Mental Development.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Monica Ibrahim, Principal investigator, Assiut University
Other Study IDs: Phenylketonuria
Record Dates: First submitted 2020-03-07; First posted 2020-03-10 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Phenylketonuria
  Interventions: Dietary Supplement: phenylalanine restricted diet
- normal healthy children
  Interventions: Dietary Supplement: phenylalanine restricted diet

INTERVENTIONS:
Dietary Supplement: phenylalanine restricted diet — Infants with hyperphenylalaninemia on special formula and diet

SUMMARY:
The study aim is to follow up body growth(body weight by kg, length by cm, head circumference, abdominal circumference, and body mass index ) and mental development of infants on phenylalanine restricted diet in comparison with normal matchable infants.

DETAILED DESCRIPTION:
Phenylketonuria is rare genetic disease caused by mutation in gene of phenylalanine (Phe) hydroxylase that converts Phenylalanine into tyrosine. The absence of this enzyme leads to elevation and accumulation of Phenylalanine and, increased phenylketones in urine (hence PKU), and also leads to decrease myelin formation, dopamine, norepinephrine, and serotonin production.

Phenylketonuria worldwide affects about 1 in 12,000 babies.

In Egypt the incidence rate reported 1 : 3000 (0.03%), The actual prevalence of PKU in this study were 1/3000. This is higher than that reported by Temtamy25, who found in a pilot study on 15,000 newborns in 3 governorates in Egypt that the incidence of PKU was 1/ 7500 . The latest consensus in Egypt showed that at least one million babies are born every year.

Phenylalanine hydroxylase deficiency (PAH deficiency) causes a spectrum of disorders, including classic phenylketonuria (PKU).

A rarer form of hyperphenylalaninemia is tetrahydrobiopterin deficiency, which occurs when the PAH enzyme is normal, and a defect is found in the biosynthesis or recycling of the cofactor tetrahydrobiopterin (BH4).

Elevations of phenylalanine in the plasma depend on the degree of enzyme deficiency. In patients with severe PAH deficiency (previously referred to classic phenylketonuria ), plasma phenylalanine levels on unrestricted diet usually exceed 20 mg/dL (>1,200 μmol/L). In affected infants with plasma concentrations >20 mg/dL, excess phenylalanine is metabolized to phenylketones (phenylpyruvate and phenylacetate) that are excreted in the urine, giving rise to the term phenylketonuria (PKU).

If left untreated and not detected early , irreversible damage may occur due to the accumulation of Phenylalanine and its metabolites in the body and will affect the growth and development of patients .

Without treatment most children develop profound and irreversible intellectual disability, seizures, hyperactive behavior with autistic features, psychiatric symptoms, eczema, musty body odor, and light pigmentation.

Newborn screening is performed to detect the disease and initiate treatment before any damage is done. The blood sample is usually taken by heel prick, typically performed 2-7 days after birth. This test can reveal elevated phenylalanine levels after one or two days of normal infant feeding. PKU is commonly included in the newborn screening panel of many countries and Egypt , with varied detection techniques. Most babies are screened for PKU soon after birth.

If left untreated and not detected early , irreversible damage may occur due to the accumulation of Phenylalanine and its metabolites in the body and will affect the growth and development of patients .

Without treatment most children develop profound and irreversible intellectual disability, seizures, hyperactive behavior with autistic features, psychiatric symptoms, eczema, musty body odor and light pigmentation.

Newborn screening is performed to detect the disease and initiate treatment before any damage is done. The blood sample is usually taken by heel prick, typically performed 2-7 days after birth. This test can reveal elevated phenylalanine levels after one or two days of normal infant feeding. PKU is commonly included in the newborn screening panel of many countries and Egypt , with varied detection techniques. Most babies are screened for PKU soon after birth.

Treatment is with a diet low in foods that contain phenylalanine and special supplements. Babies should use a special formula with a small amount of breast milk. The diet should begin as soon as possible after birth and be continued for life. People who are diagnosed early and maintain a strict diet can have normal health and a normal life .

The target of the treatment is to reach optimal health ranges of phenylalanine (or "target ranges") are between 120 and 360 µmol/L or equivalently 2 to 6 mg/dL, and aimed to be achieved during at least the first 10 years, to allow the brain to develop normally.

The dietary restriction in phenylketonuria should be only in protein diet (phenylalanine),while fat and carbohydrate diet don't need to be restricted.

Lifelong treatment will provide the best effect on growth and development, prevents neurocognitive impairment and abnormal executive functioning and helps maintaining mental health.

Anthropometric measures are important for evaluating the growth development and nutritional status of infants with phenylketonuria.

The dietary restriction in phenylketonuria should be only in protein diet (phenylalanine),while fat and carbohydrate diet don't need to be restricted.

Lifelong treatment will provide the best effect on growth and development, prevents neurocognitive impairment and abnormal executive functioning and helps maintaining mental health.

Anthropometric measures are important for evaluating the growth development and nutritional status of infants with phenylketonuria.

Intelligence and mental development in PKU PKU results, in untreated patients, a profound intellectual disability and more subtle cognitive deficits in individuals who were treated early and continuously. The assessment of intellectual functioning in PKU has been an important target outcome variable since the implementation of neonatal PKU screening programs in the 1960s . Research on intellectual functioning in individuals with PKU has played a significant role in guiding treatment recommendations and improving outcomes.

Brumm and Grant conducted a literature review examining the relationship between intellectual outcome and treatment parameters including initiation of treatment, duration of treatment, and blood phenylalanine (Phe) levels from infancy through adulthood. While current PKU treatment practices have eliminated severe neurological and cognitive impairment, evidence suggests that intellectual functioning, although typically within the average range when PKU is treated early and continuously, may not be maximized under the current definition of well-controlled PKU, which is based on blood Phe levels.

ELIGIBILITY:
Inclusion Criteria:

1. Infants with hyperphenylalaninemia on special formula and diet
2. Infants of both sexes
3. Age since birth till three years
4. Type of feeding : diet restriction of phenylalanine
5. Controls: normal healthy children match with cases in the same social class, age and sex

Exclusion Criteria:

1. Age greater than three years
2. Patients diagnosed with PKU and not regular in feeding for special diet and formula.
3. PKU patients not diagnosed since birth

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cases:Infants with hyperphenylalaninemia on special formula and diet Controls: normal healthy children match with cases in the same social class, age and sex
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Normal growth in early dietary treated patients with Phenylketonuria to assessed by body mass index in kg/m^2 | one year
  Normal growth in early dietary treated patients with Phenylketonuria to assessed by body mass index in kg/m^2
Normal growth in Early dietary treated patients with Phenylketonuria to assessed by head circumference in centimeters | one year
  Normal growth in Early dietary treated patients with Phenylketonuria to assessed by head circumference in centimeters
Normal growth in Early dietary treated patients with Phenylketonuria to assessed by abdominal circumference in centimeters | one year
  Normal growth in Early dietary treated patients with Phenylketonuria to assessed by abdominal circumference in centimeters
Mental development in early dietary treated patients with Phenylketonuria to assessed by using Emerging Pattern Of Behavior of infants | one year
  Mental development in early dietary treated patients with Phenylketonuria to assessed by using Emerging Pattern Of Behavior of infants
Comparison between early dietary treated patients with Phenylketonuria with normal matchable infants regarding normal growth and mental development | one year
  Comparison between early dietary treated patients with Phenylketonuria with normal matchable infants regarding normal growth and mental development

CONTACTS AND LOCATIONS:
Overall Officials: Farouk Hassanein, Study Director — Assiut University

REFERENCES:
- [Background] Belanger-Quintana A, Martinez-Pardo M. Physical development in patients with phenylketonuria on dietary treatment: a retrospective study. Mol Genet Metab. 2011 Dec;104(4):480-4. doi: 10.1016/j.ymgme.2011.08.002. Epub 2011 Aug 10. PMID 21878401
- [Background] Blau N. Genetics of Phenylketonuria: Then and Now. Hum Mutat. 2016 Jun;37(6):508-15. doi: 10.1002/humu.22980. Epub 2016 Mar 18. PMID 26919687
- [Background] Brumm VL, Grant ML. The role of intelligence in phenylketonuria: a review of research and management. Mol Genet Metab. 2010;99 Suppl 1:S18-21. doi: 10.1016/j.ymgme.2009.10.015. PMID 20123465
- [Background] Burgard P. Development of intelligence in early treated phenylketonuria. Eur J Pediatr. 2000 Oct;159 Suppl 2:S74-9. doi: 10.1007/pl00014388. PMID 11043149
- [Background] Cleary M, Trefz F, Muntau AC, Feillet F, van Spronsen FJ, Burlina A, Belanger-Quintana A, Gizewska M, Gasteyger C, Bettiol E, Blau N, MacDonald A. Fluctuations in phenylalanine concentrations in phenylketonuria: a review of possible relationships with outcomes. Mol Genet Metab. 2013 Dec;110(4):418-23. doi: 10.1016/j.ymgme.2013.09.001. Epub 2013 Sep 9. PMID 24090706
- [Background] Evans S, Daly A, MacDonald J, Pinto A, MacDonald A. Fifteen years of using a second stage protein substitute for weaning in phenylketonuria: a retrospective study. J Hum Nutr Diet. 2018 Jun;31(3):349-356. doi: 10.1111/jhn.12510. Epub 2017 Sep 21. PMID 28940742
- [Background] Evans S, Daly A, MacDonald J, Preece MA, Santra S, Vijay S, Chakrapani A, MacDonald A. The micronutrient status of patients with phenylketonuria on dietary treatment: an ongoing challenge. Ann Nutr Metab. 2014;65(1):42-8. doi: 10.1159/000363391. Epub 2014 Sep 4. PMID 25196394
- [Background] Jani R, Coakley K, Douglas T, Singh R. Protein intake and physical activity are associated with body composition in individuals with phenylalanine hydroxylase deficiency. Mol Genet Metab. 2017 Jun;121(2):104-110. doi: 10.1016/j.ymgme.2017.04.012. Epub 2017 Apr 28. PMID 28465125
- [Background] Dokoupil K, Gokmen-Ozel H, Lammardo AM, Motzfeldt K, Robert M, Rocha JC, van Rijn M, Ahring K, Belanger-Quintana A, MacDonald A. Optimising growth in phenylketonuria: current state of the clinical evidence base. Clin Nutr. 2012 Feb;31(1):16-21. doi: 10.1016/j.clnu.2011.09.001. Epub 2011 Sep 29. PMID 21959353
- [Background] MacDonald A, Gokmen-Ozel H, van Rijn M, Burgard P. The reality of dietary compliance in the management of phenylketonuria. J Inherit Metab Dis. 2010 Dec;33(6):665-70. doi: 10.1007/s10545-010-9073-y. Epub 2010 Apr 7. PMID 20373144
- [Background] Meli C, Bianca S. Dietary control of phenylketonuria. Lancet. 2002 Dec 21-28;360(9350):2075-6. doi: 10.1016/S0140-6736(02)11958-1. No abstract available. PMID 12504428
- [Background] Mitchell JJ, Trakadis YJ, Scriver CR. Phenylalanine hydroxylase deficiency. Genet Med. 2011 Aug;13(8):697-707. doi: 10.1097/GIM.0b013e3182141b48. PMID 21555948
- [Background] Rocha JC, van Rijn M, van Dam E, Ahring K, Belanger-Quintana A, Dokoupil K, Gokmen Ozel H, Lammardo AM, Robert M, Heidenborg C, MacDonald A. Weight Management in Phenylketonuria: What Should Be Monitored. Ann Nutr Metab. 2016;68(1):60-5. doi: 10.1159/000442304. Epub 2015 Nov 25. PMID 26598928